CLINICAL TRIAL: NCT01760811
Title: CETUXIMAB Given for 3 Weeks as Neoadjuvant Treatment Followed by 6 Weeks of Cetuximab+RT Post Surgery in Locally Advanced Squamous Cell Carcinoma of the Tongue ; A NEW PARADIGM OF TREATMENT
Brief Title: CETUXIMAB Given for 3 Weeks as Neoadjuvant Treatment in Locally Advanced Tongue Cancer ; A NEW PARADIGM OF TREATMENT
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Collaborators: Kaplan Medical Center (Other); Meir Medical Center (Other)
Responsible Party: Principal Investigator, popovtzer aron, Head of head and neck cancer unit, Rabin Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RMC0766
Record Dates: First submitted 2013-01-02; First posted 2013-01-04 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Squamous Cell Carcinoma
Keywords: tongue; Squamous cell carcinoma; locally advanced; cetuximab
MeSH Terms: conditions — Carcinoma, Squamous Cell | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cetuximab ,neoadjuvant administration (Other): Drug administration ,Cetuximab(merck Serono )given neoadjuvant ,3 courses prior surgery followed by post operatve radiation and Cetuximab
  Interventions: Drug: Erbitux,merck serono

INTERVENTIONS:
Drug: Erbitux,merck serono — cetuximab loading dosage 400mg/m2 followed by weekly 250mg/m2 2 weeks

SUMMARY:
To compare the Disease free survival (DFS) rate of a preoperative cetuximab treatment followed by operation and postoperative radiation-cisplatin-cetuximab treatment paradigm for advanced oral cavity cancer, , with the DFS rate of historical controls (from the RTOG 9501 and EORTC 22931 studies in which treatment was with surgery followed by radiotherapy and cisplatin) with a similar stage of the disease.

DETAILED DESCRIPTION:
This non-randomized, open-label, single center phase II study, will determine if patients with advanced oral tongue cancer that are treated with induction doses of cetuximab followed by treatment with radiation therapy concurrently with cetuximab and cisplatin (when indicated by positive margins or extra-capsular extension), will have improved PFS and improved survival and feasible toxicity, compared with patients treated in previous clinical trials (RTOG 9501 and EORTC 22931) with standard therapy: radiotherapy of 60 Gy with or without a 6-Gy boost (RTOG 9501) or 66 Gy (EORTC 22931) delivered through a conventional fractionation regimen of five once-daily sessions per week, and cisplatin in a dose of 100 mg/m2 on days 1, 22, and 43.. Twenty five patients will be recruited. Cetuximab treatment will be started (day 0) with 400 mg/m2 followed by two doses of 250 mg/m2 (once weekly on day 7 and 14). Surgery will be performed on day 31 followed by treatment with radiation therapy concurrently with cetuximab (250 mg/m2, once weekly) and cisplatin 35 mg/m2 (days 70-112; when indicated by positive margins or lymph nodes with extra-capsular extension). PET-CT and biopsies will be performed before starting with cetuximab, just before surgery and after chemo-cetuximab-RT to determine efficacy of treatment, and to compare the diagnostic properties of the PET-CT with that of the biopsies. The changes, before and after treatment with cetuximab, of protein levels in saliva, and tumor tissue and of microRNA levels in tumor tissue will be studied and correlated with PFS. The quality of life will be assessed. Data from clinical trials RTOG 9501 and EORTC 22931 will be used as historical controls.

ELIGIBILITY:
Inclusion Criteria:

Pathologically confirmed, previously untreated, resectable squamous cell carcinoma of the tongue at disease stage III or IV; Age ≥18 to ≤80; Eastern Cooperative Oncology Group (ECOG) Performance status 0-1;willingto give written informed consent for participation in this study -

Exclusion Criteria:

Any prior head and neck malignancy or other malignancy in the last 5 years but BCC; Prior head and neck radiation; Documented evidence of distant metastases; Pregnancy or lactation; Clinically significant cardiovascular disease; Known hypersensitivity to any of the components of the treatment; Legal incapacity; Clinically relevant neuropathy; Any medical or psychiatric illness which would compromise the patient's ability to tolerate this treatment, or interfere with the study objectives. -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
PROGRESSION FREE SURVIVAL | 2 YEARS
  : To compare the Disease free survival (DFS) rate of a preoperative cetuximab treatment followed by operation and postoperative radiation-cisplatin-cetuximab treatment paradigm for advanced oral cavity cancer, , with the DFS rate of historical controls (from the RTOG 9501 and EORTC 22931 studies in which treatment was with surgery followed by radiotherapy and cisplatin) with a similar stage of the disease

SECONDARY OUTCOMES:
Adverse event rate | 2 years
  To evaluate the frequency and severity of adverse events (AEs) for this treatment paradigm.
Biomarker prediction | 2 years
  To evaluate the correlation between changes in expression levels of several biomarkers related to cell apoptosis and tumor progression: the endothelial growth factor receptor pathway, p53, human papilloma virus, BCL-2, BCL-X(L), and acid ceramidase - before and after treatment - with survival rates, PFS and response rates

OTHER OUTCOMES:
Micro -RNA | 2 YEARS
  To evaluate the role of downregulation of microRNAs according to the outcome of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Aron Popovtzer, MD, Principal Investigator — Tel Aviv University
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel